CLINICAL TRIAL: NCT05254431
Title: The Effect of Interval Exercise on Functional Outcomes in Veterans With COPD and OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E3535-W; 1IK2RX003535 (NIH)
Record Dates: First submitted 2022-01-28; First posted 2022-02-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: COPD; OSA
Keywords: COPD; OSA; Overlap Syndrome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise trial of 12 weeks moderate intensity interval exercise in Veterans with COPD and OSA that compares exercise group to standard of care control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): The Experimental Design is a randomized trial of Moderate intensity interval training (5-minute intervals at 50% VO2peak 3 times weekly for 12 weeks) in Veterans with COPD and OSA compared with standard of care controls
  Interventions: Behavioral: Exercise
- Usual Care (No Intervention): Participants in the control group will be instructed to maintain their routine activity level for 12 weeks

INTERVENTIONS:
Behavioral: Exercise — Novel Moderate Intensity Interval Exercise
  The Experimental Design is a randomized trial of moderate intensity interval training (5-minute intervals at 50% VO2peak 3 times weekly for 12 weeks) in Veterans with COPD and OSA compared with standard of care controls
  Other Names: MIIT
  Arms: Exercise

SUMMARY:
The term "Overlap Syndrome" (OS) is used to describe the presence of both chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) in a single patient. Due to premature aging, patients with OS are prone to developing functional decline up to 20 years earlier than the general population. The International Classification of Functioning, Disability and Health (ICF) evaluates functional status in chronic pulmonary disease globally in 5 domains. The investigators propose to study validated outcomes in 3 of these domains: 1) participation in life situations; 2) physical activity; and 3) cardiovascular health. The investigators long-term goal is to develop an exercise strategy tailored to Veterans with OS which will reduce the risk of functional decline through increased PA.

DETAILED DESCRIPTION:
The term "Overlap Syndrome" (OS) is used to describe the presence of both chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) in a single patient. Veterans with OS who also have excessive daytime sleepiness (EDS-OS) are at highest risk for functional decline yet have the greatest barriers to exercise training. Thus, there is a critical need to identify novel exercise strategies that meet the individual needs and capacities of Veterans with EDS-OS. The investigators propose to test moderate intensity interval training (MIIT), a novel exercise intervention whose translation into durable lifestyle change may be facilitated by the feasibility of short bouts of increased PA. The investigators proposal addresses key knowledge gaps in rehabilitation research by investigating the clinical phenotype of EDS-OS to determine the association with functional outcomes and response to a novel exercise intervention with the goal to reduce functional decline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD and OSA, i.e., Overlap Syndrome Diagnosis of Overlap Syndrome (both COPD and OSA), confirmed in CPRS from spirometry or pulmonary function test of FEV1/FVC <70 for COPD and a polysomnogram or home-based study for OSA.
* Montreal Cognitive Assessment (MoCA) >20

Exclusion Criteria:

* CAD, as defined by anyone of the following: history of CABG, prior positive stress test for ischemia, infarction or angina or medical problem
* Orthopedic problems as defined by joint pain limiting ambulation
* Fall risk, defined as more than 2 falls in the prior month
* Hospitalization in prior month
* Daytime home oxygen 6. Participation in structured exercise, defined by the Physical Activity Scale for the Elderly (PASE) as more than 1 hour of activity spent in moderate activity and any strenuous activity performed over prior 7 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Scale number on Epworth Sleepiness Scale | 12 weeks
  Change from baseline ESS at 12 weeks ESS is daytime sleepiness scale, lower numbers better Scale goes from 0- not sleepy at all; to 20 -very sleepy
Number of Daily Steps | 12 weeks
  Change from baseline in Daily Steps at 12 weeks All participants will wear a wrist accelerometer (ActiGraph wGT3X-BT) for 7 days at baseline and the end of intervention phase to record daily steps. ActiLife software will be used to run validation algorithms and calculate mean daily steps.
Concentration of Serum hs-CRP (mg/dL) | 12 weeks
  Change from baseline in Serum hs-CRP (mg/dL) at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Madalina Macrea, MD PhD, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (1):
- Salem VA Medical Center, Salem, VA, Salem, Virginia, United States

IPD SHARING:
Plan to Share IPD: No